CLINICAL TRIAL: NCT01460355
Title: Surgery Associated to Intraoperative Botulinum Toxin A for Large Angle Horizontal Strabismus: a Pilot Study
Brief Title: Comparison of Two Treatments for Strabismus Correction: Botulinum Toxin A Associated to Surgery and Surgery Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Nilza Minguini, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unicamp-CEP- 427/2006
Record Dates: First submitted 2011-10-16; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Esotropia; Exotropia
Keywords: strabismus surgery; botulinum toxin; esotropia; exotropia; blepharoptosis
MeSH Terms: conditions — Esotropia; Exotropia; Blepharoptosis | interventions — Botulinum Toxins, Type A; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin plus surgery (Active Comparator): Intraoperative injection of 5U (0.1 ml) of Botulinum Toxin will be given to the recessed muscle during surgery
  Interventions: Drug: Botulinum Toxin Type A
- Saline solution plus surgery (Placebo Comparator): Saline solution (0,1 ml)will be given to the recessed muscle during surgery procedure
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Botulinum Toxin Type A — injection of 5U in 0.1ml of saline solution will be given to the recessed muscle
  Other Names: BTA
  Arms: Botulinum toxin plus surgery
Drug: saline solution — injection of 0,1ml of saline solution will be given to the recessed muscle
  Other Names: saline
  Arms: Saline solution plus surgery

SUMMARY:
Two different treatments were given to large angle horizontal strabismus (eso and exotropia) adult patients who agree to participate of the study. Inform consents were required for participants. Group 1 (12 patients) received conventional recess-resect surgery plus intraoperative injection of botulinum toxin A (5U). Group 2 (11 patients) received only conventional recess-resect surgery. The patients were randomly located in one of the groups. The angles of horizontal deviation were compared between the groups before and six months after treatment.

DETAILED DESCRIPTION:
Patients underwent recess/resection surgery on the non-fixating eye using conventional technique under local anesthesia. The extent of surgery was determined based on our usual amounts. Before re-attaching the recessed muscle to the sclera, 5 units of botulinum toxin in 0.1 ml of hyaline solution were, or 0.1 ml of hyaline solution alone were was injected into the posterior muscle belly by the surgeon who was unaware of the contents of each syringe.

ELIGIBILITY:
Inclusion Criteria:

* adults with large angle horizontal strabismus

Exclusion Criteria:

* oblique muscle disfunction
* previous strabismus surgery
* dissociated vertical deviation
* paretic or restrictive deviation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
percentage of decrease of the initial angle of strabismus | 6 to 12 months
  The percentages of decrease of the initial angle of strabismus were accessed by subtracting the final deviation of the initial deviation, dividing the result by the initial deviation and multiplying it by 100.

SECONDARY OUTCOMES:
frequency of induced blepharoptosis | From the first to the last post operative day of follow up
  The presence of induced blepharoptosis was detected by simple inspection and was reported as positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Nilza Minguini, MD, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- State University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Owens PL, Strominger MB, Rubin PA, Veronneau-Troutman S. Large-angle exotropia corrected by intraoperative botulinum toxin A and monocular recession resection surgery. J AAPOS. 1998 Jun;2(3):144-6. doi: 10.1016/s1091-8531(98)90004-0. PMID 10532749
- [Background] Khan AO. Two horizontal rectus eye muscle surgery combined with botulinum toxin for the treatment of very large angle esotropia. A pilot study. Binocul Vis Strabismus Q. 2005;20(1):15-20. PMID 15828866
- [Background] Ozkan SB, Topaloglu A, Aydin S. The role of botulinum toxin A in augmentation of the effect of recession and/or resection surgery. J AAPOS. 2006 Apr;10(2):124-7. doi: 10.1016/j.jaapos.2005.11.011. PMID 16678746
- See also: The page shows the summaries of Unicamp Theses on Botulinum Toxin — http://www.bibliotecadigital.unicamp.br